CLINICAL TRIAL: NCT07147101
Title: A Prospective, Non-interventional Study of Different First-line Immunotherapy in Advanced Hepatocellular Carcinoma Patients: Efficacy and Immune Microenvironment Dynamics
Brief Title: Different First-line Immunotherapy for Advancer Hepatocellular Carcinoma: A Prospective Observational Study on Efficacy and Immune Microenvironment
Acronym: HCC-IM-1
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, professor, Fudan University
Other Study IDs: HCC-IM-1
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — sintilimab; camrelizumab; apatinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A baseline tumor biopsy and blood collection before initiation of treatment, followed by a second tumor biopsy with paired blood collection after the first response evaluation will be planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCC cohort 1: Sintilimab plus bevacizumab biosimilar
  Interventions: Drug: Sintilimab; Drug: Bevacizumab Biosimilar
- HCC cohort 2: Camrelizumab plus Rivoceranib
  Interventions: Drug: Camrelizumab; Drug: Rivoceranib
- HCC cohort 3: O+Y
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be administered by IV, 200 mg every 3 weeks
  Groups: HCC cohort 1: Sintilimab plus bevacizumab biosimilar
Drug: Bevacizumab Biosimilar — Bevacizumab biosimilar will be administered by IV, 15 mg/kg every 3 weeks.
  Groups: HCC cohort 1: Sintilimab plus bevacizumab biosimilar
Drug: Camrelizumab — Camrelizumab will be administered by IV, 200 mg every 2 weeks.
  Groups: HCC cohort 2: Camrelizumab plus Rivoceranib
Drug: Rivoceranib — Rivoceranib will be administered by oral 250 mg once daily.
  Groups: HCC cohort 2: Camrelizumab plus Rivoceranib
Drug: Nivolumab — Nivolumab will be administered by IV, 1 mg/kg every 3 weeks for up to four doses, followed by nivolumab 480 mg every 4 weeks
  Groups: HCC cohort 3: O+Y
Drug: Ipilimumab — Ipilimumab will be administered by IV, 3mg/kg every 3 weeks for up to four doses.
  Groups: HCC cohort 3: O+Y

SUMMARY:
To evaluate the efficacy and immune microenvironment changes in advanced hepatocellular carcinoma (HCC) patients receiving different first-line immunotherapy.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational study evaluating the efficacy and immune microenvironment changes in advanced hepatocellular carcinoma (HCC) patients receiving different first-line immunotherapy, including anti-PD1+anti-VEGF, anti-PD1+TKI and anti-PD1+anti-CTLA4. The primary endpoint is objective response rate (ORR), with secondary endpoints including disease control rate (DCR), duration of response (DOR), time to response (TTR), progression-free survival (PFS), overall survival (OS), and immune profiling of tumor tissue and peripheral blood before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of study entry.
* Barcelona Clinic Liver Cancer stage C, or stage B not amenable to curative or locoregional therapies.
* HCC conﬁrmed by radiology, histology or cytology.
* No prior systemic therapy for HCC.
* At least one measurable site of disease as defined by RECIST1.1criteria with spiral CT scan or MRI.
* Child-Pugh scores 5-7, performance status (PS) ≤ 2 (ECOG scale).
* Adequate organ function:

  * ANC ≥1.5 × 10⁹/L, platelets ≥100 × 10⁹/L, hemoglobin ≥9 g/dL.
  * Total bilirubin ≤1.5 × ULN, AST/ALT ≤3 × ULN (≤5 × ULN if liver metastases).
  * Creatinine ≤1.5 × ULN or CrCl ≥60 mL/min.
* Willing to provide archival/fresh tumor tissue and peripheral blood samples.
* Signed informed consent.

Exclusion Criteria:

* Prior systemic therapy for HCC
* Active autoimmune disease requiring immunosuppression.
* Active infection requiring IV antibiotics.
* HIV-positive or active HBV/HCV infection (HBsAg+ with HBV DNA ≥2000 IU/mL; HCV RNA+).
* Symptomatic CNS metastases.
* Pregnancy/lactation.
* Any condition compromising protocol compliance or data interpretation per investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced hepatocellular carcinoma planed to receive first-line immunotherapy.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD).
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Time to Response (TTR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  TTR is defined as the time from the start of treatment until the first objective observation of a response (either partial response, PR, or complete response, CR), provided that the response is subsequently confirmed.
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first)
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 42 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.
Translational study | max 24 months
  Proportion of different immune cell types in tumors and blood based on RNA sequencing between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No